CLINICAL TRIAL: NCT00641017
Title: A Phase I Study of the Safety and Immunogenicity of the Recombinant Live-Attenuated Human Parainfluenza Type 1 Virus Vaccine, rHPIV1 84/del170/942A, Lot PIV1 #104A, Delivered as Nose Drops to Adults 18 to 49 Years of Age, HPIV1-Seropositive Children 15 to 59 Months of Age, and HPIV1-Seronegative Infants and Children 6 to 59 Months of Age
Brief Title: Safety of and Immune Response to Recombinant Live-Attenuated Parainfluenza Type 1 Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 248
Record Dates: First submitted 2008-03-05; First posted 2008-03-21 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Parainfluenza; Virus Diseases
MeSH Terms: conditions — Paramyxoviridae Infections; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 and 2 - Adults (Experimental): One immunization of 1x10^6 TCID50 rHPIV1 84/del170/942A administered intranasally via nose drops at study entry
  Interventions: Biological: rHPIV1 84/del170/942A, Lot PIV1 #104A vaccine
- 3A - Seropositive Children (Experimental): One immunization of 1x10^6 TCID50 rHPIV1 84/del170/942A administered intranasally via nose drops at study entry
  Interventions: Biological: rHPIV1 84/del170/942A, Lot PIV1 #104A vaccine
- 3B - Seropositive Children (Placebo Comparator): One dose of 1x10^6 TCID50 rHPIV1 84/del170/942A placebo administered intranasally via nose drops at study entry
  Interventions: Biological: Placebo
- 4A - Seronegative Infants and Children (Experimental): One immunization of 1x10^5 TCID50 rHPIV1 84/del170/942A administered intranasally via nose drops at study entry
  Interventions: Biological: rHPIV1 84/del170/942A, Lot PIV1 #104A vaccine
- 4B - Seronegative Infants and Children (Placebo Comparator): One dose of 1x10^5 TCID50 rHPIV1 84/del170/942A placebo administered intranasally via nose drops at study entry
  Interventions: Biological: Placebo
- 5A - Seronegative Infants and Children (Experimental): One immunization of 1x10^6 TCID50 rHPIV1 84/del170/942A administered intranasally via nose drops at study entry
  Interventions: Biological: rHPIV1 84/del170/942A, Lot PIV1 #104A vaccine
- 5B - Seronegative Infants and Children (Placebo Comparator): One dose of rHPIV1 84/del170/942A placebo administered intranasally via nose drops at study entry
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rHPIV1 84/del170/942A, Lot PIV1 #104A vaccine — Live attenuated Human Parainfluenza Type 1 Virus Vaccine
  Arms: 1 and 2 - Adults; 3A - Seropositive Children; 4A - Seronegative Infants and Children; 5A - Seronegative Infants and Children
Biological: Placebo — Placebo for rHPIVI1 84/del170/942A, Lot PIV1 #104A vaccine
  Arms: 3B - Seropositive Children; 4B - Seronegative Infants and Children; 5B - Seronegative Infants and Children

SUMMARY:
Human Parainfluenza Virus Type 1 (HPIV1) is a leading cause of viral respiratory infections in children, the elderly, and those with compromised immune systems. HPIV1 is also the leading cause of viral croup in children under 6 years old. The purpose of this study is to determine the safety of and immune response to a HPIV1 vaccine, rHPIVI1 84/del170/942A, in 2 groups of adults and then in children who have been previously exposed to HPIV1. Once the safety of this vaccine has been established in these groups, an additional 2 groups of infants and children who have not been previously exposed to HPIV1 will be vaccinated. Naïve infants and children are the most vulnerable to naturally circulating HPIV1 and are the target population of this vaccine.

DETAILED DESCRIPTION:
HPIV1 infection can result in severe respiratory illness that often leads to the hospitalization of infants and young children. HPIV1 is responsible for approximately 6% of all pediatric hospitalizations for respiratory tract diseases and is a main cause of severe lower respiratory tract diseases, including pneumonia and bronchiolitis in children less than 6 years old. The purpose of this study is to determine the safety of and immune response to a HPIV1 vaccine, rHPIVI1 84/del170/942A, in 5 main volunteer group: first in adults (group 1 and 2), and then in seropositive children (group 3). The last 2 groups will be seronegative infants and children that are split into 2 dosing groups; one group of seronegative infants and children will receive a lower dose of vaccine (group 4) and a second group of seronegative infants and children (group 5) will receive a higher dose of vaccine. This study will last approximately 8 weeks per group. Additional information about each of the groups is as follows:

Groups 1 and 2 will consist of 35 adults total, 18 to 49 years of age. These groups will receive one immunization with rHPIV1 84/del170/942A at study entry. Immunization will be given as nose drops. Study visits will occur on Days 3, 4, 5, 6, 7, 10, and 28. Medical history, vital signs, clinical assessment, and nasal wash will occur at most visits. Blood and urine tests will occur at selected visits. A urine pregnancy test will occur for females at study entry. Follow-up phone reports will also be required on Day 56.

Enrollment into Group 3 will begin only after safety data from Groups 1 and 2 are evaluated. Group 3 will consist of 15 seropositive children, 15 to 59 months of age. This group will receive either one immunization of rHPIV1 84/del170/942A or placebo at study entry. Immunization will be given as nose drops. Study visits will occur on Days 3, 4, 5, 6, 7, 10, and 28. Medical history, vital signs, clinical assessment, and nasal wash will occur at most visits. Blood and urine tests will occur at selected visits. Parents will be required to submit reports over the phone throughout the study. These reports will include the temporal temperature from the previous day.

Enrollment into Group 4 will begin only after safety data from Group 3 are evaluated. Group 4 will consist of 21-30 seronegative infants and children, 6 to 59 months of age. This group will receive either one immunization of rHPIV1 84/del170/942A or placebo at study entry. Immunization will be given as nose drops. Study visits will occur on Days 3, 5, 7, 10, 12, 14, 17, 19, 21, 28, and 56. Medical history, vital signs, clinical assessment, and nasal wash will occur at most visits. Blood tests will occur at selected visits. Parents will be required to submit reports over the phone throughout the study. These reports will include the temporal temperature from the previous day.

Enrollment into Group 5 will begin only after safety data from Group 4 are evaluated. Group 5 will consist of 21-30 seronegative infants and children 6 to 59 months of age. This group will receive either one immunization of rHPIV1 84/del170/942A or placebo at study entry. The immunization will be given as nose drops. The vaccine dosage that participants receive in Group 5 will be greater than the dose in Group 4. Study visits will occur on Days 3, 5, 7, 10, 12, 14, 17, 19, 21, 28, and 56. Medical history, vital signs, clinical assessment, and nasal wash will occur at most visits. Blood tests will occur at selected visits. Parents will be required to submit reports over the phone throughout the study. These reports will include the temporal temperature from the previous day.

ELIGIBILITY:
Adult Inclusion Criteria:

* In good health
* Available for the duration of the trial
* Available for post-inoculation telephone contact
* For females, must agree to use effective birth control methods for the duration of the study

Seropositive Children Inclusion Criteria:

* In good health
* Seropositive for HPIV1
* Available for the duration of the study

Seronegative Infants and Children Inclusion Criteria:

* In good health
* Seronegative for HPIV1 antibody
* Available for the duration of the study

Adult Exclusion Criteria:

* Neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease
* Condition, in the opinion of the investigator, that will not allow the participant to comply with the protocol
* Alcohol or drug abuse
* History of anaphylaxis
* History of splenectomy
* Diagnosis of asthma within 2 years of study entry
* HIV-infected
* Hepatitis C infection
* Hepatitis B infection
* Abnormal urinalysis
* Known immunodeficiency syndrome
* Current use of nasal or systemic steroid medications
* Receipt of blood products within 3 months of study entry
* Current smoker unwilling to stop smoking for the duration of the study. The decision to exclude a potential subject is made by the investigator based upon the potential subject's medical history and physical examination.
* Participation in another investigational vaccine or drug trial within 30 days of receiving the investigational vaccine
* Receipt of live vaccine within 4 weeks or a killed vaccine within 2 weeks or immune globin within 3 months prior to receiving the investigational vaccine
* Previous immunization with an HPIV1 vaccine
* Known hypersensitivity to any vaccine component
* Participants whose profession and/or personal responsibilities involve caring for children less than 6 months of age or for immunosuppressed individuals
* Persistent systolic blood pressure more than 140 mm Hg or diastolic pressure more than 90 mm Hg
* Body mass index (BMI) more than 35
* Pregnant or breastfeeding

Seropositive and Seronegative Infants and Children Exclusion Criteria:

* Known or suspected impairment of immunological functions as determined by the investigator
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with HPIV1 vaccine
* Current use of nasal or systemic steroid medications
* Previous serious vaccine-associated adverse event or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including reactive airway disease as determined by the investigator
* Member of household that includes an immunocompromised individual or infant less than 6 months of age
* Attends day care with infants less than 6 months of age or immunosuppressed individuals. More information about this criterion can be found in the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of receiving the investigational vaccine or while study is occurring

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2008-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reaction events and other adverse events in each cohort | Throughout study
Amount of vaccine virus shed by each participant | Throughout study
Amount of serum antibody and mucosal antibody induced by the vaccine in each participant | Throughout study

SECONDARY OUTCOMES:
Phenotypic stability of vaccine virus shed | Throughout study
Number of vaccinated children and infants infected with rHPIV1 | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bartlett EJ, Amaro-Carambot E, Surman SR, Collins PL, Murphy BR, Skiadopoulos MH. Introducing point and deletion mutations into the P/C gene of human parainfluenza virus type 1 (HPIV1) by reverse genetics generates attenuated and efficacious vaccine candidates. Vaccine. 2006 Mar 24;24(14):2674-84. doi: 10.1016/j.vaccine.2005.10.047. Epub 2005 Nov 15. PMID 16364511
- [Background] Bartlett EJ, Castano A, Surman SR, Collins PL, Skiadopoulos MH, Murphy BR. Attenuation and efficacy of human parainfluenza virus type 1 (HPIV1) vaccine candidates containing stabilized mutations in the P/C and L genes. Virol J. 2007 Jul 2;4:67. doi: 10.1186/1743-422X-4-67. PMID 17605811
- [Derived] Karron RA, San Mateo J, Thumar B, Schaap-Nutt A, Buchholz UJ, Schmidt AC, Bartlett EJ, Murphy BR, Collins PL. Evaluation of a Live-Attenuated Human Parainfluenza Type 1 Vaccine in Adults and Children. J Pediatric Infect Dis Soc. 2015 Dec;4(4):e143-6. doi: 10.1093/jpids/piu104. Epub 2014 Nov 12. PMID 26582883